CLINICAL TRIAL: NCT00278187
Title: Phase II Open-Label Study of Volociximab (M200) in Combination With Erlotinib (Tarceva™) in Previously Treated Patients With Locally Advanced (Stage IIIb) or Metastatic (Stage IV) Non-Small Cell Lung Cancer
Brief Title: Volociximab and Erlotinib in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453542; UCLA-0504066-01; PDL-M200-1206
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-02

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — volociximab; Erlotinib Hydrochloride

INTERVENTIONS:
Biological: volociximab
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Monoclonal antibodies, such as volociximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Volociximab may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving volociximab together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving volociximab together with erlotinib works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the response rate in patients with locally advanced (stage IIIB) or metastatic (stage IV) non-small cell lung cancer treated with volociximab and erlotinib hydrochloride.

Secondary

* Evaluate the time to disease progression and duration of response in patients treated with this regimen.
* Evaluate the safety of this drug regimen in these patients.
* Evaluate the pharmacokinetics this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive volociximab IV over 30 minutes once every 2 weeks and oral erlotinib hydrochloride daily for 52 weeks in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed at 3 and 6 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced (stage IIIB) or metastatic (stage IV) non-small cell lung cancer (NSCLC)
* Failed ≥ 1 prior chemotherapy regimen OR refused first-line therapy
* Measurable disease
* No active and untreated CNS tumor or metastasis

  * Previously treated CNS tumor(s) allowed if CT scan or MRI shows clear-cut response or resolution of the original lesion(s)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Hemoglobin ≥ 9.0 g/dL
* WBC ≥ 2,500/mm^3
* Absolute neutrophil count ≥ 1,000/mm^3 (growth factor independent)
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN) (5 times ULN if patient has liver metastases)
* Alkaline phosphatase ≤ 5 times ULN
* Serum creatinine ≤ 2.0 mg/dL
* PT/PTT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective (double barrier or abstinence) contraception
* No uncontrolled seizure disorder or active neurological disease
* No thromboembolic events (i.e., stroke or deep vein thrombosis) within the past year
* No clinically significant medical condition that would complicate compliance with study treatment or be exacerbated by bleeding, including but not limited to:

  * Known bleeding disorders, such as coagulation defects and thrombasthenias
  * Active gastric or duodenal ulcer
  * History of gastrointestinal (GI) bleeding requiring transfusion within the past year
  * History of tumor bleeding
  * History of significant hemoptysis requiring intervention (i.e., transfusion, laser therapy, surgical treatment, or radiation) within the past year
* No known active infections requiring IV antibiotics, antivirals, or antifungals (e.g., HIV, hepatitis B, or hepatitis C infection)
* No unstable cardiac disease, including any of the following:

  * Poorly controlled angina
  * Congestive heart failure
  * Arrhythmias
  * Myocardial infarction within the past year
  * Acute ischemia by ECG
  * Untreated significant conduction abnormality

    * Bifascicular block (defined as left anterior hemiblock in the presence of right bundle branch block)
    * Second- or third-degree atrioventricular block
* No asthma or oxygen-dependent chronic pulmonary disease
* No cerebrovascular event (e.g., stroke or transient ischemic attack) within the past year
* No peripheral vascular disease requiring surgery within the past year
* No clinically significant or unstable medical condition, including, but not limited to, any of the following:

  * Diabetes mellitus requiring insulin
  * Uncontrolled hypertension
  * Uncontrolled or symptomatic orthostatic hypertension
* No serious psychiatric illness, active alcoholism, or drug addiction that may preclude study treatment
* No condition that, in the investigator's opinion, would make the patient unsuitable for study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior immunotherapy, including monoclonal antibodies, or vaccine therapy allowed
* No systemic biologic, immunotherapy, or radiation therapy within the past 4 weeks

  * Local radiotherapy to a single site of bone metastasis within the past 2 weeks allowed provided patient has recovered from any side effects
* No prior volociximab, epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors, or inhibitors of α5β1 integrin (antibodies or small molecules)
* No known hypersensitivity to murine proteins or chimeric antibodies or other components of study drugs
* No other investigational drug within the past 4 weeks or 5 half-lives (whichever is longer)
* No monoclonal antibody therapy within the past 4 weeks or 5 half-lives (whichever is longer)
* No major surgery (e.g., thoracotomy) within 4 weeks prior to study entry
* No minor surgery (e.g., central venous line placement) within 1 week prior to study entry
* No sargramostim (GM-CSF) or filgrastim (G-CSF) within the past 7 days
* No prior bone marrow or stem cell transplantation
* No concurrent chronic medications that would interfere with study drug assessment including, but not limited to:

  * High-dose glucocorticoids (prednisone ≥ 20 mg/day or equivalent)
  * Chronic nonsteroidal anti-inflammatory drugs (NSAIDs)

    * Infrequent or as occasion requires use of NSAIDs allowed
* No concurrent high-dose aspirin (> 81 mg/day), high-dose warfarin, or heparin

  * Aspirin ≤ 81 mg/day, low-dose warfarin (1 mg/day), or low-dose heparin for IV-catheter patency allowed
* No concurrent chemotherapy, therapeutic radiation, or anticancer hormonal therapy
* No other concurrent immunotherapy
* No other concurrent potentially antiangiogenic therapy (e.g., cyclo-oxygenase-2 inhibitors, thalidomide, or tretinoin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-07

PRIMARY OUTCOMES:
Proportion of patients with confirmed tumor response

SECONDARY OUTCOMES:
Time to disease progression
Duration of response
Adverse events and serious adverse events
Pharmacokinetics
Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Figlin, MD, FACP, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States